CLINICAL TRIAL: NCT07135167
Title: Compassionate Use Study of Epi-ON Corneal Collagen Crosslinking Performed Using UVA Exposure on Eyes With Ectatic Corneal Diseases for Subjects With Down Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Woolfson Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEI-CXL-002
Record Dates: First submitted 2025-08-05; First posted 2025-08-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome (DS); Keratoconus; Pellucid Marginal Degeneration; Forme Fruste Keratoconus (FFK)
Keywords: corneal crosslinking (CXL); cornea; riboflavin; vitamin B2; ultraviolet
MeSH Terms: conditions — Down Syndrome; Keratoconus; Corneal Diseases | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Enrolled and treated subject arm (Experimental): Epi-ON corneal cross-linking (CXL)
  Interventions: Combination Product: Epi-ON corneal cross-linking (CXL)

INTERVENTIONS:
Combination Product: Epi-ON corneal cross-linking (CXL) — Corneal cross-linking involves the following steps:
  * applying riboflavin (Vitamin B2 eye drops) to the eye, then
  * exposing the eye to ultraviolet (UV-A) light for 20 minutes.

SUMMARY:
The goal of this clinical trial is to study the effects of an experimental (not Food and Drug Administration (FDA)-approved) treatment called corneal crosslinking (CXL) for conditions in which the cornea becomes progressively thin, steep, and misshapen, causing vision to be blurred.

CXL is performed by putting riboflavin (vitamin B2) drops onto the eye and then exposing it to ultraviolet (UVA) light at about the same intensity as you get outdoors on a bright, sunny day. It is designed to stop the progression of disease by strengthening the cornea. Study participants will be 8 years of age or older and have a diagnosis of Down syndrome.

The main question it aims to answer is:

* Does CXL help prevent or slow the progression of someone's corneal condition and vision loss?

Participants will:

* Attend up to a total of 7 in office visits over the course of 6 months, where several eye and vision tests will be given.

Receive CXL (applying riboflavin (Vitamin B2 eye drops) to the eye, then exposing the eye to ultraviolet (UV-A) light for 20 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 8 years of age or older, male or female, of any race.
2. Have a diagnosis of Down syndrome or other cognitive, developmental, or medical conditions that precludes the subject from reliably following instructions or performing some of the study examination procedures.
3. Have a diagnosis of keratoconus, pellucid marginal degeneration, progressive ectasia after previous CXL treatment, other ectatic condition, or forme fruste keratoconus based on topography, tomography, and slit lamp examination.
4. Provide written informed consent and a signed HIPAA form. Pediatric subjects less than 14 years of age must sign an assent, and a parent or legal guardian must sign an informed consent. If the subject has impaired consent capacity, determined by the consenter, the consent form must be signed by the subject's legally authorized representative on behalf of the subject.
5. Satisfactory completion of the standardized clinical decision tool evaluation of patient suitability for CXL. (See Section 7.2.3)
6. Be willing and able to follow all instructions to the best of his/her abilities and comply with the schedule for follow-up visits.

Exclusion Criteria:

1. Normal corneal topography.
2. A history of previous corneal transplant in the study eye.
3. Minimum corneal thickness < 300 (measured by Pentacam and Ultrasound) at the screening exam.
4. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye to future complications or prevent the possibility of improved vision, for example:

   1. History of, or active, corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
   2. Clinically significant corneal scarring in the central cornea that, in the investigator's opinion, will not allow the subject to achieve functional vision, even with contact lens correction, after the crosslinking procedure.
5. A known contraindication, sensitivity, or allergy to the test article or its components or to study medications.
6. Nystagmus or any other condition that would prevent a steady gaze during the crosslinking treatment or other diagnostic tests.
7. If female, pregnant, lactating or planning a pregnancy, or having a positive urine pregnancy test prior to the randomization of, or treatment of either eye during the course of the study. [NOTE: If female and capable of becoming pregnant, must agree to use a medically acceptable form of birth control for at least one week prior to the treatment visit and to continue one month following treatment. ]

7. Inability to remove soft or scleral contact lenses at least 3 days before initial and follow-up examinations.

8. Inability to remove rigid gas-permeable contact lenses at least 2 weeks before initial and follow-up examinations.

9. Inability to return for required postoperative examinations. 10. Presence or history or any other condition or finding that, in the investigator's opinion, makes the subject unsuitable as a candidate for crosslinking or study participation or may confound the outcome of the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures for efficacy is corneal curvature, as measured by Kmax with the Pentacam, in the treated eyes. | From enrollment to the end of treatment at 6 months.
  Primarily using measurements to assess improvement of vision.
Improvement of vision as assessed by corrected distance visual acuity (CDVA). | From enrollment to the end of treatment at 6 months.
  Change in CDVA compared to the baseline examination will be evaluated at 6 months postoperatively. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.

SECONDARY OUTCOMES:
Improvement in vision as measured by high order aberrations (HOA). | From enrollment until end of follow-up period at 6 months.
  At the Sponsor-Investigator's discretion, the change in HOA from baseline may be evaluated at 6 months postoperatively for the eyes that underwent preoperative and postoperative wavefront testing. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.
Improvement in vision as assessed by change in coma. | Enrollment through the follow-up phase at 6 months.
  At the Sponsor-Investigator's discretion, the change in coma from baseline may be evaluated at 6 months postoperatively for the eyes that underwent preoperative and postoperative wavefront testing. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.
Improved vision as assessed by Uncorrected Visual Acuity (UCVA). | Enrollment through the end of the follow-up period at 6 months.
  Change in UCVA compared to the baseline examination will be evaluated at 6 months postoperatively. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Woolfson Eye Institute, Atlanta, Georgia
  - Woolfson Eye Institute, Canton, Georgia
  - Woolfson Eye Institute, Cumming, Georgia
  - Woolfson Eye Institute, Douglasville, Georgia
  - Woolfson Eye Institute, Lawrenceville, Georgia
  - Woolfson Eye Institute, Marietta, Georgia
  - Woolfson Eye Institute, Snellville, Georgia
  - Woolfson Eye Institute, Asheville, North Carolina
  - Woolfson Eye Institute, Chattanooga, Tennessee
  - Woolfson Eye Institute, Johnson City, Tennessee
  - Woolfson Eye Institute, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided